CLINICAL TRIAL: NCT07388940
Title: Pilot Study of MammoGRIP for Breast Positioning, Image Quality, and Patient Comfort in Mammography
Acronym: MammoGRIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: E-25-145
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Mammography
Keywords: Mammogram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MammoGRIP (Experimental): MammoGRIP® is an FDA-cleared, single-use, topical foam adhesive solution designed to improve technologist grip during breast positioning for mammography. In this study, MammoGRIP® will be used in accordance with the manufacturer's instructions and applied immediately before positioning each breast for imaging.
  Interventions: Device: MammoGRIP

INTERVENTIONS:
Device: MammoGRIP — MammoGRIP® is an FDA-cleared, single-use, topical foam adhesive solution designed to improve technologist grip during breast positioning for mammography. In this study, MammoGRIP® will be used in accordance with the manufacturer's instructions and applied immediately before positioning each breast for imaging.

SUMMARY:
To evaluate the effectiveness of MammoGRIP® in improving mammographic image quality and minimizing repeated breast positioning compared to standard practice without MammoGRIP®.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-75 years undergoing routine screening or diagnostic mammography
* Ability to provide informed consent
* Prior mammogram results are available for the patient in Epic

Exclusion Criteria:

* History of bilateral mastectomy
* Active skin condition or open wounds on the breast or chest
* Known allergy to components of MammoGRIP®

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Image quality | Images from the current scan will be compared to the images from a historical scan (1 year prior)
  - Pectoralis muscle visualization in MLO and or CC views
Image Quality | Images from the current scan will be compared to the images from a historical scan (1 year prior)
  Nipple in profile
Image quality | Images from the current scan will be compared to the images from a historical scan (1 year prior)
  Visualization of the inframammary fold
Image Quality | Images from the current scan will be compared to the images from a historical scan (1 year prior)
  Lack of skin folds
Image Quality | Images from the current scan will be compared to the images from a historical scan (1 year prior)
  Distance from the chest wall to the nipple on MLO and CC views (less than 1cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Hospital, Englewood, New Jersey, United States